CLINICAL TRIAL: NCT01838343
Title: Efficacy of Ultrasound to Guide Management During a Rapid Response Event
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 218-12
Record Dates: First submitted 2013-04-05; First posted 2013-04-24 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Hemodynamic Instability; Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Ultrasound (No Intervention): Patients randomized to no ultrasound will get standard diagnostic and therapeutic interventions that are clinically indicated during the rapid response event.
- Ultrasound (Experimental): Patients randomized to ultrasound will get a goal-directed ultrasound performed by a critical care fellow along with standard diagnostic and therapeutic interventions that are clinically indicated during the rapid response event.
  Interventions: Other: Ultrasound

INTERVENTIONS:
Other: Ultrasound — Goal-directed ultrasound using a GE Vscan performed by a critical care fellow trained in ultrasonography.
  Other Names: Ultrasound to be performed by GE Vscan.
  Arms: Ultrasound

SUMMARY:
Rapid response team systems have been implemented in numerous hospitals throughout the world with the goal of improving the identification and safety of hospitalized patients who are clinically deteriorating. Despite their theoretical benefit, rapid response systems have not been proven in the medical literature to ultimately change outcomes.

The traditional physical exam is helpful in evaluating and treating unstable medical patients during these types of events but has significant limitations of deceased sensitivity and specificity of findings. Ultrasound is a known tool for more accurately assessing patients in shock and respiratory failure in the ICU by highly trained operators but to the investigators knowledge has not been studied in the setting of rapid response events on hospital wards by critical care fellows after focused training. The investigators aim to assess the impact of ultrasound performed by critical care fellows during rapid response events.

DETAILED DESCRIPTION:
This is an randomized controlled trial to determine if portable critical care ultrasound use is feasible, if its findings change clinical decision making by critical care fellows and whether ultrasound can improve patient outcomes during rapid response events at Beth Israel Medical Center.

Patients for whom a rapid response has been called for cardiac or respiratory failure will be randomized to either have a bedside ultrasound performed by a critical care fellow at the time of rapid response or to undergo a bedside ultrasound only if clinically indicated and specifically requested by the RRT leader.

For all patients on whom a rapid response is called with shock or respiratory failure who are randomized to the intervention group, a designated ultrasound critical care fellow will document their ranked top 2 preliminary cause for either shock or respiratory failure on a data collection instrument (DCI). These clinical (i.e. pre-ultrasound) diagnoses will be based on history, physical exam and all ancillary testing available prior to ultrasound performance. Available ancillary testing will be documented.

An ultrasound exam will then be performed by the designated ultrasound fellow using a portable hand-carried unit (GE Vscan) and the findings documented on the same DCI. The GE Vscan will be used for all ultrasounds performed during this study. The ultrasound study will take approximately 5 -10 minutes and will not interfere with alternative evaluation or treatment modalities deemed to be necessary during the rapid response.

The critical care ultrasound fellow will then provide the RRT leader team with their 2 most likely post ultrasound diagnosis for shock and respiratory failure and then document these on the DCI. Any changes to management made as a result of the ultrasound exam, including all new ancillary tests and therapeutic interventions will be recorded.

At 72 hours following the initial event the ICU or general medical attending physician will be asked to document the "final" diagnosis as to the cause of the initial shock or respiratory failure. This "final" diagnosis will serve as the "gold standard" to allow the assessment of accuracy of the pre-ultrasound and post-ultrasound diagnoses.

Patients randomized to the standard care group will not have an ultrasound performed at the time of rapid response unless it is deemed medically necessary by the responding RRT leader or critical care fellow. This is the current practice approach at the investigators hospital where ultrasound is performed only when clinically indicated.

The study investigators will obtain all DCI's as well as the final diagnosis from the attending physician at 72 hours, and will enter this data into a database that will not contain any unique patient identifiers.

The patient's time in respiratory failure and time in shock will be recorded as primary outcome measures. Secondary outcomes of in-hospital mortality, utilization of CT scan and chest x-ray in the 24 hours following rapid response and hospital length of stay will also be recorded. Also measured will be variability in pre and post-ultrasound diagnosis as well as changes in management following ultrasound performance.

ELIGIBILITY:
Inclusion Criteria: Patients for whom a rapid response is called who have:

1. Hemodynamic instability as defined by:

   * Systolic blood pressure less than 90 mmHg or less than 40 mmHg from previously established baseline
   * Heart rate greater than 130 beats per minute
   * Known elevated lactate above normal value.
2. Hypercapnic or hypoxemic respiratory failure as judged by the responding critical care fellow.

Exclusion Criteria: Patients for whom a rapid response has been called who:

1. Are not hemodynamically unstable and not in respiratory failure.
2. Are hemodynamically unstable but who have an obvious source of bleeding to explain hemodynamic instability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Time in shock | Immediately after rapid response
  Time on vasopressors following the rapid response event and for 8 weeks thereafter.
Time in respiratory failure | From immediately after rapid response event and for 8 weeks thereafter.
  Time period that the patient requires invasive or non-invasive mechanical ventilation.

SECONDARY OUTCOMES:
Mortality | During hospitaliztion or for 8 weeks thereafter.
  Death during the hospitalization that the rapid response occured during.
Diagnosis variation following ultrasound | Immediately after ultrasound and for 1 day thereafter.
  Agreement between pre-ultrasound and post-ultrasound diagnosis.
Utilization of chest x-ray | Following rapid response event and one day thereafter.
  Frequency of chest x-ray performance will be measured during the 24 hours immediately following the rapid response event.
Utilization of CT scan | Following rapid response event for one day thereafter.
  Frequency of CT scan performance will be measured during the 24 hours immediately following the rapid response event.
Length of stay | Following rapid response event and for 8 weeks thereafter.
  Hospital length of stay following rapid response event.
Management changes following ultrasound performance | Immediately following ultrasound and for one day thereafter.
  Pre-ultrasound and post-ultrasound management will be documented.

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Medical Center, New York, New York, United States